CLINICAL TRIAL: NCT06499714
Title: HighCycle Study: Effect of High Altitude on Acute Mountain Sickness in Women Related to Their Menstrual Cycle Phase: A Prospective Cohort Study at 3600 m
Brief Title: HighCycle Study: Effect of High Altitude on Acute Mountain Sickness in Women Related to Their Menstrual Cycle Phase
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); University Hospital Heidelberg (Other); Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Other Study IDs: HighCycle_AMS_MCP
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Acute Mountain Sickness
Keywords: Women; Hypoxia; Prevention; Acetazolamide; Altitude
MeSH Terms: conditions — Altitude Sickness; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women in luteal MCP: Women being in their luteal MCP on the day of ascent to high altitude.
  Interventions: Other: Exposure to 3600 m
- Women in follicular MCP: Women being in their follicular MCP on the day of ascent to high altitude.
  Interventions: Other: Exposure to 3600 m

INTERVENTIONS:
Other: Exposure to 3600 m — Participants will travel to and stay for 2 days at an altitude of 3600 m.

SUMMARY:
Prospective cohort study investigating the menstrual cycle phase (MCP)-dependent incidence of acute mountain sickness (AMS) in women travelling to 3600 m.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking women, age 18-44 years, without any disease and need of regular medication (including oral contraceptives).
* BMI >18 kg/m2 and <30 kg/m2
* Born, raised and currently living at altitudes <1000 m
* Written informed consent
* Premenopausal, eumenorrheic cycle

Exclusion Criteria:

* Other types of contraceptives (hormonal intrauterine device, vaginal ring, subcutaneous injections or implants, among others)
* Pregnancy or nursing
* Anaemic (haemoglobin concentration <10g/dl)
* Any altitude trip <4 weks before the study
* Allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, non-smoking, premenopausal women, age 18-44 years, without any disease and need of regular medication (including oral contraceptives).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Mountain Sickness (AMS) Incidence, LLS 2018 | Day 1 to 3 at 3600 m
  MCP-related difference in the AMS incidence. AMS incidence will be defined as a Lake Louise Questionnaire version 2018 score of ≥3.

SECONDARY OUTCOMES:
Acute Mountain Sickness (AMS) Incidence, LLS 1993 | Day 1 to 3 at 3600 m
  MCP-related difference in the AMS incidence. AMS incidence will be defined as a Lake Louise Questionnaire version 1993 score of ≥3.
Acute Mountain Sickness (AMS) Severity, LLS 2018 | Day 1 to 3 at 3600 m
  MCP-related difference on the AMS severity assessed by the Lake Louise Questionnaire version 2018.
Acute Mountain Sickness (AMS) Severity, LLS 1993 | Day 1 to 3 at 3600 m
  MCP-related difference on the AMS severity assessed by the Lake Louise Questionnaire version 1993.
Arterial blood gases | Day 2 at 760 m and day 2 at 3600 m
  MCP-related difference on the arterial blood gases (pH, PaO2, PaCO2, SaO2).
Hypoxic ventilatory response | Day 2 at 760 m
  MCP-related difference in the hypoxic ventilatory response assessed under FiO2 of 0.115 and while cycling on a bicycle at 30% of predicted maximal work capacity.
Perceived pain visualization | Day 1 to 3 at 3600 m
  MCP-related difference on perceived pain sensations, visualized by the SMaRT tablet app

CONTACTS AND LOCATIONS:
Overall Officials: Michael Furian, Prof. Dr., Study Chair — University of Zurich; Talant Sooronbaev, Prof. Dr., Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Gorod Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided